CLINICAL TRIAL: NCT05497323
Title: Effectivity and Safety of Combination Cream of Salicylic Acid, Aqua Posae Filiformis, Niacinamide, Lipohydroxy Acid, Procerad and Zinc PCA as Adjuvant Therapy for Acne Vulgaris Mild to Moderate
Brief Title: Effectivity and Safety of Combination Cream of Salicylic Acid, Aqua Posae Filiformis, Niacinamide, Lipohydroxy Acid, Procerad and Zinc PCA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Dr. dr. Irma Bernadette S. Sitohang, SpKK(K) - Head of Cosmetic Dermatology Division of Dermatology and Venereology Department of Faculty of Medicine Universitas Indonesia / Cipto Mangunkusumo Hospital, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EffectivityCombiAquaPosae
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
Keywords: combination cream; aqua posae; adjuvant therapy
MeSH Terms: conditions — Acne Vulgaris | interventions — Lidocaine, Prilocaine Drug Combination; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Cream Group (Experimental): Group 2 will use Adapalene 0.1% cream intermittently every two nights and the combination cream every morning. Group 3 will use Adapalene 0.1% cream every night and the combination cream every morning. Subjects were evaluated on day 28 and day 56.
  Interventions: Drug: Combination Cream
- Adapalene 0,1% cream (Other): The control group (Group 1) will use Adapalene 0.1% cream only every night. Subjects were evaluated on day 28 and day 56.
  Interventions: Drug: Adapalene 0,1% cream

INTERVENTIONS:
Drug: Combination Cream — The combination cream consists of Salicylic Acid, Aqua Posae Filiformis, Niacinamide, Lipohydroxy Acid, Procerad and Zinc PCA, were applied every morning by group 2 and group 3.
  Other Names: La Roche Posay, Effaclar Duo (+), dermocosmetic
  Arms: Combination Cream Group
Drug: Adapalene 0,1% cream — Adapalene 0,1 % cream were given to subjects to be applied every night in group 1 and group 3, and intermittently every two nights in group 2.
  Other Names: Evalen®, topical acne agents
  Arms: Adapalene 0,1% cream

SUMMARY:
This clinical study will compare the effectivity and safety of combination cream of Salicylic Acid, Aqua Posae Filiformis, Niacinamide, Lipohydroxy Acid, Procerad, and Zinc PCA as adjuvant therapy for acne vulgaris patients. These combination cream will be tested by mild to moderate acne vulgaris patients. Participants will be female patients aged 15-50 years old and divided into three groups. The control group (Group 1) will use Adapalene 0.1% cream only every night. Group 2 will use Adapalene 0.1% cream intermittently every two nights and the combination cream every morning. Group 3 will use Adapalene 0.1% cream every night and the combination cream every morning.

DETAILED DESCRIPTION:
This study is an experimental study with a randomized controlled trial (RCT) design on mild to moderate acne vulgaris patients who met the inclusion criteria. This study will be conducted in five Dermatology and Venereology Education Centers in Indonesia located in Jakarta (Rumah Sakit Umum Pusat Nasional dr. Cipto Mangunkusumo), Jakarta (Rumah Sakit Pusat Angkatan Darat Gatot Soebroto), Padang (Rumah Sakit Umum Pusat Dr. M. Djamil), Surakarta (Rumah Sakit Umum Daerah Dr. Moewardi), and Malang (Rumah Sakit Umum Daerah Dr. Saiful Anwar). Group 1 as control group, will receive Adapalene 0.1% cream only every night. Group 2 will receive Adapalene 0.1% cream only intermittently every two nights, and the combination cream every morning. Group 3 will use Adapalene 0.1% cream every night and the combination cream every morning. All participants will be evaluated in day 28 and 56. Therapy evaluation will be assessed based on the Global Acne Severity Scale (GEA Score), Indonesia Acne Expert Meeting (IAEM Score), Level of Seborrhoea, Clinician Erythema Assessment Scale (CEA), facial skin analysis with Janus Skin Facial Analysis, and evaluation of the quality of life using Cardiff Acne Disability Index and Acne-Quality of Life (Acne-QoL) specifically for participants aged older than 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 15 - 50 years
* Mild and moderate acne vulgaris according to IAEM and GEA.
* Patients are willing to participate in the study until it is finished.

Exclusion Criteria:

* History of allergy to dermatocosmetic products.
* Undergoing other acne therapy, medication, or invasive action in the last month.
* Pregnant or breastfeeding patients

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 284 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of acne severity | re-evaluation on day 28 and day 56 of therapy
  Based on Global Acne Severity Scale (GEA Score). On a scale of 0-5, 0 indicates almost no lesions, while 5 indicates severe acne.
Change of acne severity | re-evaluation on day 28 and day 56 of therapy
  Based on Indonesia Acne Expert Meeting (IAEM score). The scale consists of mild, moderate, and severe.
Change of Level Of Seborrhea | re-evaluation on day 28 and day 56 of therapy
  The level of seborrhea is assessed subjectively by participants on a scale of 0 (minimum level) - 10 (maximum level)
Change of erythema | re-evaluation on day 28 and day 56 of therapy
  Based on Clinician Erythema Assessment Scale (CEA) to assess the degree and extent of erythema. The scale ranges from 0-5; 0 indicates no erythema, while 4 indicates severe erythema.
Change of quality of life | re-evaluation on day 28 and day 56 of therapy
  Assessed using Cardiff Acne Disability Index. Cardiff Acne Disability Index questionnaire is an instrument to measure the quality of life of acne vulgaris patients. This instrument has 5 self-answered questions by the patient (for subjects aged≥ 18 years).
Change of quality of life | re-evaluation on day 28 and day 56 of therapy
  Assessed using Acne-Quality of Life. Acne-QoL is an instrument consisting of 19 questions divided into 4 categories: self-perception, social relationships, emotional effects, and acne symptoms. The total score of Acne-QoL is 0-114. The higher total score for each category obtained will interpret that the quality of life of acne vulgaris patients is getting better.
Facial Analysis Examination With Janus Facial Analysis System | re-evaluation on day 28 and day 56 of therapy
  Assessed using the Janus Facial Analysis System®. Janus Facial Analysis System will issue data related to the patient's facial condition.

CONTACTS AND LOCATIONS:
Overall Officials: Irma BS Sitohang, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Lilik Norawati, MD, Study Director — Departemen Ilmu Kesehatan Kulit dan Kelamin Rumah Sakit Pusat Angkatan Darat Gatot Soebroto,; Satya WY Yenny, MD, Study Director — Departemen Ilmu Kesehatan Kulit dan Kelamin Rumah Sakit Umum Pusat Dr. M. Djamil, Padang; Arie Kusumawardani, Study Director — Departemen Ilmu Kesehatan Kulit dan Kelamin Rumah Sakit Umum Daerah Dr. Moewardi, Surakarta; Sinta Murlistyarini, Study Director — Departemen Ilmu Kesehatan Kulit dan Kelamin Rumah Sakit Umum Daerah Saiful Anwar, Malang
Locations (5):
- Indonesia (5):
  - Rumah Sakit Umum Daerah Dr. Moewardi, Surakarta, Central Java
  - Rumah Sakit Pusat Angkatan Darat Gatot Soebroto, Jakarta, DKI Jakarta
  - Rumah Sakit Umum Pusat Cipto Mangunkusumo, Jakarta, DKI Jakarta
  - Rumah Sakit Umum Daerah Saiful Anwar, Malang, East Java
  - Rumah Sakit Umum Pusat Dr. M. Djamil, Padang, West Sumatra